CLINICAL TRIAL: NCT05980234
Title: PMCF Study to Provide Safety, Performance, and Clinical Benefits Data of the Longevity IT Oblique and Offset Liners in Primary and Revision Total Hip Arthroplasty - A Retrospective Enrollment/Prospective Follow-up Consecutive Series Study
Brief Title: MDR - Longevity IT Oblique and Offset Liners
Status: Terminated | Type: Observational
Why Stopped: Zimmer Biomet received the CE mark for the Continuum and Trilogy IT Acetabular System, which includes the Longevity IT Offset and Oblique Liners, in June 2024.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-107H
Record Dates: First submitted 2023-07-24; First posted 2023-08-07 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Non-inflammatory Degenerative Joint Disease (NIDJD); Avascular Necrosis; Protrusio Acetabuli; Traumatic Arthritis; Slipped Capital Femoral Epiphyses; Fracture of the Pelvis; Diastrophic Variant; Osteoarthritis; Fused Hip
MeSH Terms: conditions — Osteonecrosis; Slipped Capital Femoral Epiphyses; Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Longevity IT Oblique Liners: The Longevity IT Oblique liner was designed to provide variable joint anteversion and abduction.
  Interventions: Device: Total Hip Arthroplasty with Longevity IT Oblique Liners
- Longevity IT Offset Liners: The Longevity IT Offset liner was designed to lateralize the center of rotation of the cup.
  Interventions: Device: Total Hip Arthroplasty with Longevity IT Offset Liners

INTERVENTIONS:
Device: Total Hip Arthroplasty with Longevity IT Oblique Liners — Primary or Revision Total Hip Arthroplasty using the Longevity IT Oblique liners according to the approved indications and compatible device.
  Groups: Longevity IT Oblique Liners
Device: Total Hip Arthroplasty with Longevity IT Offset Liners — Primary or Revision Total Hip Arthroplasty using the Longevity IT Offset liners according to the approved indications and compatible device.
  Groups: Longevity IT Offset Liners

SUMMARY:
The objective of this retrospective enrollment/prospective follow-up consecutive series PMCF study is to collect data confirming safety, performance, and clinical benefits of the Longevity IT Oblique and Offset liners when used for primary or revision total hip arthroplasty (implants and instrumentation) at a minimum of 10-year follow-up.

DETAILED DESCRIPTION:
The objective of this retrospective enrollment/prospective follow-up consecutive series PMCF study is to collect data confirming safety, performance, and clinical benefits of the Longevity IT Oblique and Offset liners when used for primary and revision total hip arthroplasty (implants and instrumentation) at 1, 3, 5, 7, and 10 years*. The subject devices have been on the market since 2010 but have insufficient data to support 10 years of clinical history. A prospective aspect to the study will be utilized to collect long-term data.

ELIGIBILITY:
Inclusion Criteria:

* Study devices must have been implanted following the appropriate surgical technique and IFU
* Patient must be 18 years of age or older
* Patient must be willing and able to sign or verbally consent using the IRB approved informed consent
* Patient must have undergone primary or revision hip arthroplasty with the Longevity IT Oblique and/or Offset liners according to a cleared indication, which includes the following:
* Noninflammatory degenerative joint disease including osteoarthritis and avascular necrosis, protrusio acetabuli, traumatic arthritis, slipped capital, epiphysis, fused hip, fracture of the pelvis, and diastrophic variant
* Revision where other devices or treatments have failed
* Patient must have reached full skeletal maturity

Exclusion Criteria:

* Off-label use of study devices
* Osteoradionecrosis
* Neuromuscular compromise, vascular deficiency or other conditions in the affected limb that may lead to inadequate skeletal fixation
* Systemic or local infection
* Uncooperative patient or patient with neurologic disorders who is incapable of following directions
* Patient is known to be pregnant or nursing
* Patient is a prisoner
* Patient is a known alcohol or drug abuser
* Patient has a psychiatric illness or cognitive deficit that will not allow for proper informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population should be a consecutive series of subjects implanted with the Longevity IT Oblique and/or Offset liners in either primary or revision THA. Up to 52 implanted hips with the Oblique liners and up to 52 implanted hips with the Offset liners will be included in the study.
  The study population for primary statistical analysis will be comprised of males and females who satisfy the inclusion/exclusion criteria outlined in the protocol. To avoid potential selection bias, each Investigator will offer study participation to each consecutive eligible patient presenting as a potential candidate. Eligible candidates who express interest in study participation will be offered Informed Consent.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent Adverse Events (safety) | 10 years
  This will be assessed by recording the incidence and frequency of revisions, complications, and adverse events with particular focus on those that may be related to the study device.

SECONDARY OUTCOMES:
Pain and Functional Performance - Oxford Hip Score | 10 years
  "The Oxford Hip Score is patient-reported outcome instrument which contains 12 questions on activities of daily living that assess function and residual pain in patients undergoing total hip replacement surgery.
  Grading the Oxford Hip Score 0 to 19-May indicate severe hip arthritis... 20 to 29-May indicate moderate to severe hip arthritis... 30 to 39-May indicate mild to moderate hip arthritis... 40 to 48-May indicate satisfactory joint function..." Oxford Hip Score. (n.d.) Segen's Medical Dictionary. (2011). Retrieved August 19 2022 from https://medical-dictionary.thefreedictionary.com/Oxford+Hip+Score
Performance and Clinical Benefits - Harris Hip Score | 10 years
  Patient Assessment: reported Harris Hip Score (if available)
  Harris Hip Score:
  The HHS is divided into three sections. The first section questions is about pain and its impact, which are answered by the patient or client. The second and third sections require the physiotherapist to assess the patient or client's hip joint and function.
  The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. Results can be recorded and calculated online. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Performance and Clinical Benefits - Activity Level | 10 years
  Patient Assessment: activity level
  Records patient's activity level on a 10-point scale from 'wholly inactive' to 'regularly particpates in impact sports.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No